CLINICAL TRIAL: NCT01675921
Title: Implementation of ACT Through Facebook for Teenagers With Asthma
Acronym: C2MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-P-000674/1
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma; Facebook; teenagers; ACT
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants will continue to receive medical care from their doctor as usual.
  Participants will have access to this study website at the start and at the end of the study.
- Facebook group (Experimental): Participants will continue to receive medical care from their doctor as usual.
  Participants will have access to the study website at all times throughout the study.
  Participants will have access to the secret study group on Facebook for 12 months.
  Participants will take the ACT survey once a month for 12 months.
  Interventions: Other: Facebook group

INTERVENTIONS:
Other: Facebook group — Facebook will be used to remind participants to take the ACT survey once every month for 12 months.
  Arms: Facebook group

SUMMARY:
The investigators hypothesize that at the end of the 12-month trial, teenagers regularly self-monitoring their asthma control with ACT administered through Facebook will have improved ACT scores as compared with teenagers receiving usual care.

DETAILED DESCRIPTION:
The investigators propose to administer the Asthma Control Test (ACT), a clinically validated and reliable measure of asthma control, to a pediatric pulmonary patient population, using novel channels to improve usage of the tool and health outcomes. The investigators will administer ACT to patients using Facebook to monitor asthma control and notify clinicians when there is deterioration of control.

The goal is to improve health outcomes in patients with asthma by measuring adherence to the use of monitoring tool, follow-up visits to their specialist, and hospitalization/Emergency Department (ED) visits. To achieve this, the investigators will use a novel technology platform that is simple, secure, private and easily scalable to other relevant sites and groups, without the need for additional investment. Currently, patients take the ACT survey only during their scheduled office appointments. The aim of the study is to increase the use of ACT to monitor patients who see a pediatric pulmonologist to promote regular self-monitoring.

ACT is a short symptom-based survey consisting of 5 questions, validated in English and Spanish. Participants will receive reminders on Facebook every month to login to the study website to complete the ACT survey therefore allowing patients to easily take the survey on a regular basis, and receive reminders and educational content in the media spaces they already inhabit. Participants would receive reminders and links in the same way they would receive other reminders or notifications from Facebook. The system will rate asthma control and send patients and their specialist notification of status if it reaches critical levels, defined as a score of 14 or lower on the ACT survey. This will be a system generated notification, based on a protocol developed in conjunction with the physicians at the Massachusetts General Hospital (MGH) pediatric pulmonary department.

The intervention will study the efficacy of electronic social networks in engaging teenagers in their asthma control over time, using a simple but effective symptom-based survey tool. Both patients and providers would receive notifications in case of deteriorating control, which could result in early intervention and lead to better clinical outcomes by prompting timely intervention by the clinician. The Center for Connected Health (CCH) will work with the MGH Department of Pulmonology, as well as the Pediatric Asthma group at Partners Community HealthCare Inc. (PCHI) to enroll ambulatory teenagers with asthma in the research study for one year.

120 participants will be enrolled and randomly assigned to one of two groups.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers age 14-17 years inclusive.
* Diagnosis of asthma by a PCP or a specialist at a Partners affiliated hospital/health center.
* Access to computer with internet.
* Active email account
* Fluency in English (spoken and written)
* Be on controller medications (such as: inhaled corticosteroids, cromolyn sodium and nedocromil sodium, long-acting beta-agonists (LABAs), and methylxanthines) to control asthma and prevent symptoms from developing.
* Have an active account on Facebook

Exclusion Criteria:

* Disability or co-morbidity precluding regular access to the internet.
* Cognitive impairment.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) scores | 0 to 12 months
  Assess the effect of the Facebook intervention (also referred to as "Connect 2 My ACT" intervention on trends of ACT scores in teenagers diagnosed with asthma

SECONDARY OUTCOMES:
Emergency Department (ED) visits and Hospital Admissions | 0 to 12 months
  Compare frequency of ED and hospital admissions between the intervention and control groups
Engagement | 0 to 12 months
  To assess participant engagement in the program (total number of times ACT survey taken divided by 12)
Provider engagement | 0 to 12 months
  To assess provider engagement in the program (# of times reached out to patient when alerted)
Patient engagement and Emergency Department (ED) visits | 0 to12 months
  To correlate participant engagement with change in ED visits and hospital admissions.
Satisfaction with intervention | at 12 months
  To assess usability and satisfaction with the Facebook study group by administering a survey at completion of study
Change in knowledge about asthma | 0 to12 months
  To assess changes in level of knowledge about asthma using the Asthma Self-Management Questionnaire, a standardized and validated survey instrument

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Partners Healthcare, Center for Connected Health
Locations (1):
- Partners Center for Connected Health, Boston, Massachusetts, United States